CLINICAL TRIAL: NCT05191576
Title: Sleep Problems in Epileptic Children and Their Caregivers: Associations With Psychometric
Brief Title: Sleep Problems in Epileptic Children and Their Caregivers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, İpek Dokurel, Principal Investigator, Ege University
Other Study IDs: E.148753
Record Dates: First submitted 2021-12-28; First posted 2022-01-13 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Epileptic Children,Sleep Disturbances,Maladaptive Behaviors
Keywords: Children; Epilepsy; CSHQ; SDQ; Caregiver; Sleep disturbances
MeSH Terms: conditions — Epilepsy; Parasomnias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- epileptic children: All patients were diagnosed based on the International League Against Epilepsy (ILAE) operational clinical definition criteria for epilepsy and pediatric neurologists made the diagnosis. The patients had been receiving treatment for at least one year. Epileptic patients were grouped into idiopathic generalized or self-limiting focal epilepsy syndromes according to the International League Against Epilepsy (ILAE) criteria for epileptic seizures and syndromes and guidelines for epidemiological studies for diagnosis and classification.
  Interventions: Other: Children's sleep habits questionnaire (CSHQ)
- healthy controls: healthy controls without any complaint (e.g., behavior problems, depression, or anxiety) that could interfere with sleep.
  Interventions: Other: Children's sleep habits questionnaire (CSHQ)

INTERVENTIONS:
Other: Children's sleep habits questionnaire (CSHQ) — 1. Children's Sleep Habits Questionnaire is a validated tool to screen sleep behavior in young children's assessment of pediatric sleep problems.
  2. DSM-V Level II Sleep Disturbance- Child Report. is retrospective, 8-item self-report used to assess the pure domain of sleep disturbances in children and adolescents age of 11-17 years in the past seven days.Higher scores indicate more severe sleep disorders. High scores on a particular domain might indicate significant and problematic areas for the child that may warrant further assessment.
  3. DSM -V Sleep Disturbance -Adult Report. is used to assess the pure domain of sleep disturbances in adults for the past seven days.
     SDQ).is used to screen emotional and behavioral problems in children.
  4. SDQ is used to screen emotional and behavioral problems in children.
  Other Names: Strength and difficulties questionnaire (SDQ); Diagnostic and statistical manual of mental disorders (DSM)-V Sleep Disorders Scale-Child Report; DSM-V Sleep Disorder Scale- Adult Report

SUMMARY:
The aim of this study is to investigate the frequency of sleep problems in epileptic children and their caregivers.

DETAILED DESCRIPTION:
The study instruments include two parts. First, data on socio-demographic, height, weight, the sleep duration, caregiver's level of education (Illiterate, Preliminary school, High school, University), caregiver sleep problems, and medical background were noted. Clinical data regarding epilepsy (a type of seizure, etiology, the frequency of seizures, actual and previous antiseizure medications) were collected from interviews of participants/parents and examination. Second, the psychometric assessment tools used to evaluate all participants and caregivers; Children's sleep habits questionnaire (CSHQ), strength and difficulties questionnaire (SDQ), diagnostic and statistical manual of mental disorders (DSM)-V Sleep Disorders Scale-Child Report, DSM-V Sleep Disorder Scale- Adult Report. All participants and their caregivers completed the psychometric questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of epilepsy that based on the International League Against Epilepsy (ILAE) operational clinical definition criteria for epilepsy
* must be diagnosed by pediatric neurologists
* must receive treatment for at least one year.

Exclusion Criteria:

* to have an IQ ≤80, as measured by the Wechsler Intelligence Scale for Children-Revised Form (WISC-R) or below-average academic performance documented by last year's final school grade
* to have a history of psychiatric, developmental disorder, or psychosis
* to have a history of progressive neurological disorder other than epilepsy
* to have any complaint (e.g., behavior problems, depression, or anxiety) that could interfere with sleep
* to have a caregiver who has any medical or psychiatric condition (e.g., depression or anxiety) that could interfere with sleep.

Ages: 11 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: A total of 120 patients (epileptic patients: 50, healthy controls: 70) aged 11-17 years who were attended to the pediatric neurology outpatient clinic of Ege University Medical Faculty between February and June 2020 were recruited to this observational case-control study. In the patient group, 13 patients were excluded due to incomplete questionnaires and the following exclusion criteria. In the control group, 23 children with incomplete forms and 4 children with presence of depressive or an anxiety disorder were excludedThe study cohort consisted of 80 cases. 37 were epileptic patients as study group and 43 were similar aged healthy children as control group. The control group was matched in terms of their age, gender, and caregiver educational level
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep disturbances correlation with behavioral difficulties in epileptic children | participant would be assessed at the beginning of the study
  The subscales of sleep problems would be investigated with Diagnostic and Statistical Manual of Mental Disorders (DSM) -V Level II Sleep Disturbance- Child Report,Children's Sleep Habits Questionnaire. The subscales of behavioral problems in epileptic children would be investigated with Strength and Difficulties Questionnaire.The correlation of these subscales would be correlated with statistical methods to define significant differences.

CONTACTS AND LOCATIONS:
Locations (1):
- İpek Dokurel, Izmir, Other, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
individual deidentified participant data (including data dictionaries) will be not be shared.